CLINICAL TRIAL: NCT06565741
Title: Prospective and Randomized Analysis of Endoscopic Prostate Enucleation Using Moses 2.0 Technology Versus the New Thulium Fiber Laser in Medium and Large Prostates.
Brief Title: EEAP Using Moses 2.0 Technology vs the Thulium Fiber Laser in Medium-Large Prostates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Puigvert (Other)
Responsible Party: Principal Investigator, Ivan Schwartzmann, MD, Principal Investigator, Fundacio Puigvert
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-2024-23
Record Dates: First submitted 2024-08-13; First posted 2024-08-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Prostatic Hyperplasia; Surgery; Endoscopic Anatomical Enucleation of the Prostate (EEAP)
Keywords: Medium and Large Prostates; Endoscopic Prostate Enucleation; Endoscopic anatomical enucleation of the prostate (EEAP); Holmium laser; Thulium Fiber laser; Moses 2.0 Technology
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Patients with an indication for surgery for BPH via EEAP with a prostate volume exceeding 80cc will be included in the study on a prospective basis. Surgery will be randomly assigned using MoLEP or ThuFLEP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Endoscopic Prostate Enucleation Using Moses 2.0 Technology (Active Comparator): Pulse modulation technology in Moses 2.0 applied to Holmium Laser Endoscopic Prostate (MoLEP).
  Interventions: Procedure: MoLEP
- Endoscopic Prostate Enucleation Using the New Thulium Fiber Laser (Active Comparator): Thulium Fiber laser to endoscopic prostate enucleation (ThuFLEP).
  Interventions: Procedure: ThuFLEP

INTERVENTIONS:
Procedure: MoLEP — Patients with an indication for surgery for BPH via EEAP with a prostate volume exceeding 80cc will be included in the study on a prospective basis. Surgery will be randomly assigned using MoLEP or ThuFLEP. A qualified surgeon, having completed their learning curve for endoscopic enucleation (more than 50 cases) and possessing experience with both laser types, will perform the surgical procedure.
  Other Names: Moses 2.0 Technology
  Arms: Endoscopic Prostate Enucleation Using Moses 2.0 Technology
Procedure: ThuFLEP — Patients with an indication for surgery for BPH via EEAP with a prostate volume exceeding 80cc will be included in the study on a prospective basis. Surgery will be randomly assigned using MoLEP or ThuFLEP. A qualified surgeon, having completed their learning curve for endoscopic enucleation (more than 50 cases) and possessing experience with both laser types, will perform the surgical procedure.
  Other Names: New Thulium Fiber Laser
  Arms: Endoscopic Prostate Enucleation Using the New Thulium Fiber Laser

SUMMARY:
Introduction: Endoscopic anatomical enucleation of the prostate (EEAP) with lasers has emerged as an effective and less invasive surgical option compared to traditional methods. Among the various available laser options, Holmium laser and Thulium Fiber laser have stood out as two prominent approaches for performing endoscopic prostate enucleation. These technologies have 3 showcased their effectiveness in ablating prostatic tissue and improving urinary symptoms. Nevertheless, differences in their physical properties and modes of action may impact their success rates and clinical outcomes. In our institution it is standard practice to use one laser or the other according to their availability in the operating room.

Primary Objective: To demonstrate the superiority of MoLEP over ThuFLEP in terms of enucleation efficiency.

Secondary Objectives: a) To demonstrate the non-inferiority of MoLEP compared to ThuFLEP in terms of perioperative bleeding.

b) To demonstrate the non-inferiority of MoLEP compared to ThuFLEP in terms of postoperative hospital stay.

c) To demonstrate the non-inferiority of ThuFLEP compared to ThuFLEP in terms of perioperative complications.

d) To demonstrate the non-inferiority of MoLEP compared to ThuFLEP in terms of improvement in urinary symptoms.

e) To demonstrate the non-inferiority of MoLEP compared to ThuFLEP in terms of improvement in flowmetric variables.

Study Type: Prospective, randomized, non-blind, multicentric clinical trial. Intervention: Patients with an indication for surgery for BPH via EEAP with a prostate volume exceeding 80cc will be included in the study on a prospective basis. Surgery will be randomly assigned using MoLEP or ThuFLEP. A qualified surgeon, having completed their learning curve for endoscopic enucleation (more than 50 cases) and possessing experience with both laser types, will perform the surgical procedure.

DETAILED DESCRIPTION:
Surgery and Follow-up Schedule

* Surgeries will be performed between September 2024 and September 2025.
* Initial follow-up at 3 months.
* Completion of the first phase of the study: March 2026.

Scheduled of Visits: Selection Visit, 1-Month Postoperative Visit, 3-Month Follow-up, 6-Month Follow-up, Annual Follow-up Visit (1-3 years).

Sample size calculation was done using the main outcome variable (total surgical time). Previous studies indicate that surgical time for ThuFLEP is 71.6 minutes [8]. The time for MoLEP may be at least 5 minutes less. Accepting an alpha risk of 5% and a beta risk of 20% in a two-tailed test, a total of 120 patients are needed (60 in each study group). A common standard deviation of 9 minutes change is assumed. A loss to follow-up rate of 15% has been estimated.

Randomization between the two surgery groups will be performed using the Efron procedure to balance the groups in terms of the number of subjects. The calculation will be carried out with the !RndSeq macro for SPSS Statistics. It will be conducted centrally by a person independent of the surgeon.

Statistical Analysis: For quantitative variables, measures of central tendency and dispersion will be .provided. Normality tests will be conducted using the Shapiro-Wilk test. For qualitative variables, valid percentages will be shown. Sociodemographic and clinical data, as well as the main study variables, will be compared between study groups using the Student's t-test (Mann-Whitney U test in case of non-normality). Chi-square test or Fisher's test (if any observed frequency is <5) will be used for qualitative variables. A multivariate linear regression model will be constructed to determine variables related to surgical time. Beta coefficients and 95% confidence intervals (CI) will be determined. A preliminary study will be conducted on potential confounding and interacting factors. Adjustment will be made for clinically or bibliographically relevant variables. Interaction will be tested using the likelihood ratio test. A significant difference will be accepted in all tests with a p-value <0.05. R Studio statistical package (V2.5.1) will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 40 and 90 years.
* Patients who, due to their lower urinary tract symptoms, are candidates for

BPH surgery, including:

* Obstructive urinary symptoms evaluated through IPSS with a score >7 and QoL > 2 or acute urinary reten on refractory to catheter removal.
* Obstructive urinary flow evaluated through uroflowmetry with Qmax< 15 ml/s, obstruction demonstrated by pressure/flow study, prostatic origin haematuria refractory to medical treatment, or acute urinary retention refractory to catheter removal.

  * Prostatic volume measured by transabdominal ultrasound, transrectal ultrasound, or magnetic resonance imaging of more than 80 cc.
  * Prostate-specific antigen (PSA) < 4 ng/ml, or with multiparametric prostate magnetic resonance imaging reporting PIRADS < 3 or equal to 3 with PSA density < 15%.

Exclusion Criteria:

* Diagnosis, suspicion, or history of urethral stenosis or urethral surgery.
* History of prostate surgery or pelvic radiotherapy.
* Diagnosis or suspicion of prostate cancer or urothelial cancer.
* Body mass index superior to 30.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with an indication for BPH surgery through EAEP with a prostatic volume >80cc.
Enrollment: 120 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
SURGICAL TIME | Total time of Surgery procedure
  Difference in surgical time between MoLEP and ThuFLEP in prostates larger than 80 cc.

SECONDARY OUTCOMES:
Perioperative bleeding | From date of preoperative blood test to date of control blood test postoperatively within 24 hours after surgery
  Differences in perioperative bleeding between MoLEP and ThuFLEP. Difference in haemoglobin level between preoperative blood test and control blood test postoperatively within 24 hours after surgery).
Postoperative hospital stay | From date and time of end of surgery to date and time of hospital discharge assessed up to 1 month
  Difference in postoperative hospital stay time between MoLEP and ThuFLEP. Number of days of hospitalization after surgery. Three categories will be recorded: Ambulatory (<16 hours of stay), Less than 24 hours, More than 24 hours (individual length of stay will be recorded).
Perioperative complications | From date of surgery to date of the end of follow-up 3 years
  Difference in the incidence of perioperative complications between MoLEP and ThuFLEP. All possible complications will be recorded and classified according to the Clavien- Dindo scale from date of surgery to end of study.
Urinary symptoms | From date of enrollment to date of the end of follow-up 3 years
  Difference in improvement of urinary symptoms after MoLEP compared to ThuFLEP. IPSS questionnaire will be performed in all study visits: Changes in total score and quality of life score before and after surgery will be compared between patients undergoing MoLEP and ThuFLEP.
Flowmetric variables maximum flow | From date of surgery to date of the end of follow-up 3 years
  Difference in improvement of flowmetric values after MoLEP compared to ThuFLEP. Uroflowmetry will be performed at baseline, 3 months, 6 months and annual follow-up visits: Changes in maximum flow measured in ml/s before and after surgery will be compared between patients undergoing MoLEP and ThuFLEP.
  A uroflowmetry will be considered valid if the patient reports that it is representative of their current voiding quality and if it presents a voided volume > 150 ml.
Flowmetric variables average flow | From date of surgery to date of the end of follow-up 3 years
  Difference in improvement of flowmetric values after MoLEP compared to ThuFLEP. Uroflowmetry will be performed at baseline, 3 months, 6 months and annual follow-up visits: Changes in average flow measured in ml/s before and after surgery will be compared between patients undergoing MoLEP and ThuFLEP.
  A uroflowmetry will be considered valid if the patient reports that it is representative of their current voiding quality and if it presents a voided volume > 150 ml.
Flowmetric variables post-void residual | From date of surgery to date of the end of follow-up 3 years
  Difference in improvement of flowmetric values after MoLEP compared to ThuFLEP. Uroflowmetry will be performed at baseline, 3 months, 6 months and annual follow-up visits: Changes in post-void residual measured in ml before and after surgery will be compared between patients undergoing MoLEP and ThuFLEP.
  A uroflowmetry will be considered valid if the patient reports that it is representative of their current voiding quality and if it presents a voided volume > 150 ml.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Schwartzmann Jochamowitz, MD, Principal Investigator — Fundacio Puigvert
Locations (3):
- Spain (3):
  - Fundacio Puigvert, Barcelona, BARCELONA
  - Clinic Hospital of Barcelona, Barcelona, BARCELONA
  - Hospital Univesitari de Bellvitge, L'Hospitalet de Llobregat, BARCELONA

IPD SHARING:
Plan to Share IPD: Yes
A total of two publications with study results will be made, each differing in the follow-up time. A publication of preliminary results will be made when the last patient included in the study has completed the three-month follow-up. A second publication will be made when the last included patient completes two years of follow-up.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available when the study results are published.
Access Criteria: Open

REFERENCES:
- [Background] Enikeev D, Glybochko P, Okhunov Z, Alyaev Y, Rapoport L, Tsarichenko D, Enikeev M, Sorokin N, Dymov A, Taratkin M. Retrospective Analysis of Short-Term Outcomes After Monopolar Versus Laser Endoscopic Enucleation of the Prostate: A Single Center Experience. J Endourol. 2018 May;32(5):417-423. doi: 10.1089/end.2017.0898. Epub 2018 Mar 13. PMID 29430969
- [Background] Nottingham CU, Large T, Agarwal DK, Rivera ME, Krambeck AE. Comparison of Newly Optimized Moses Technology vs Standard Holmium:YAG for Endoscopic Laser Enucleation of the Prostate. J Endourol. 2021 Sep;35(9):1393-1399. doi: 10.1089/end.2020.0996. Epub 2021 Jul 15. PMID 33813861
- [Background] Wani MM, Sriprasad S, Bhat T, Madaan S. Is Thulium laser enucleation of prostate an alternative to Holmium and TURP surgeries - A systematic review? Turk J Urol. 2020 Nov;46(6):419-426. doi: 10.5152/tud.2020.20202. Epub 2020 Oct 9. PMID 33052829
- [Background] Fraundorfer MR, Gilling PJ. Holmium:YAG laser enucleation of the prostate combined with mechanical morcellation: preliminary results. Eur Urol. 1998;33(1):69-72. doi: 10.1159/000019535. PMID 9471043
- [Background] Elmansy H, Hodhod A, Elshafei A, Noureldin YA, Mehrnoush V, Zakaria AS, Hadi RA, Fathy M, Abbas L, Kotb A, Shahrour W. Comparative analysis of MOSESTM technology versus novel thulium fiber laser (TFL) for transurethral enucleation of the prostate: A single-institutional study. Arch Ital Urol Androl. 2022 Jun 29;94(2):180-185. doi: 10.4081/aiua.2022.2.180. PMID 35775343
- [Background] Zhang Y, Yuan P, Ma D, Gao X, Wei C, Liu Z, Li R, Wang S, Liu J, Liu X. Efficacy and safety of enucleation vs. resection of prostate for treatment of benign prostatic hyperplasia: a meta-analysis of randomized controlled trials. Prostate Cancer Prostatic Dis. 2019 Dec;22(4):493-508. doi: 10.1038/s41391-019-0135-4. Epub 2019 Feb 28. PMID 30816336
- [Background] Enikeev D, Netsch C, Rapoport L, Gazimiev M, Laukhtina E, Snurnitsyna O, Alekseeva T, Becker B, Taratkin M, Glybochko P. Novel thulium fiber laser for endoscopic enucleation of the prostate: A prospective comparison with conventional transurethral resection of the prostate. Int J Urol. 2019 Dec;26(12):1138-1143. doi: 10.1111/iju.14115. Epub 2019 Sep 22. PMID 31544290